CLINICAL TRIAL: NCT06778161
Title: Clinical Research Ethic Committee of Gaziantep University
Brief Title: Comparison of Erector Spina Plane Block and Thoracic Paravertebral Block for Analgesia After Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elzem SEN (Other)
Responsible Party: Sponsor-Investigator, Elzem SEN, Assoc.Prof., University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2021/241
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Analgesia; Thoracic Surgery
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae block group (Other)
  Interventions: Procedure: nerve block
- paravertebral block group (Other)
  Interventions: Procedure: nerve block

INTERVENTIONS:
Procedure: nerve block — Nerve block for providing analgesia after thoracotomy

SUMMARY:
This study aims to compare the postoperative analgesic efficacy of ultrasound-guided erector spinae plane block (ESPB) and thoracic paravertebral block (TPVB) in patients undergoing thoracotomy. The primary outcome is the VAS scores assessed at postoperative hours 0, 3, 6, 12, and 24 for pain at rest. The secondary outcome was tramadol and morphine consumption.

DETAILED DESCRIPTION:
This study is a retrospective study conducted after obtaining approval from the Clinical Research Ethics Committee (decision no: 2021/241, dated 07/07/2021). It was carried out by reviewing the recorded data of patients who underwent thoracotomy surgery in the Department of Anesthesiology and Reanimation at Gaziantep University Faculty of Medicine Şahinbey Research and Application Hospital between October 1, 2020, and May 31, 2021. The study was conducted in accordance with the "Ethical Principles for Medical Research Involving Human Subjects" outlined in the Declaration of Helsinki published by the World Medical Association in 2013.

This study included a total of 130 patients, aged 18-75 years, with ASA physical status scores of I, II, or III, who underwent thoracotomy surgery and received ultrasound-guided ESPB or TPVB for postoperative analgesia. Written informed consent was obtained from all participants. Patients were excluded from the study if they were emergency cases, had an ASA class IV or V status, had peripheral vascular disease, were pregnant, had heart failure, were allergic to local anesthetics, or if their medical records were inaccessible.

The patients were divided into two groups of 65 individuals each, based on the type of regional analgesia administered for thoracotomy. The groups were designated as Group 1 (patients who received ESPB) and Group 2 (patients who received TPVB). Data on patients' age, gender, ASA classification, height, body weight, BMI, comorbidities, smoking status, indication for thoracotomy, thoracotomy side, duration of operation, postoperative 0th, 3rd, 6th, 12th, 24th. VAS scores, average tramadol and morphine consumption, and the presence of postoperative nausea, pruritus, and shoulder pain were collected retrospectively from medical records.

A 20-gauge peripheral venous access was provided in the operating room, and a balanced electrolyte solution was initiated at 3-5 ml/kg/hour. After completing monitoring with electrocardiography (ECG), pulse oximetry (SpO2), and non-invasive arterial pressure (mmHg), 0.03 mg/kg midazolam (Zolamid 15 mg/3 ml, VEM İlaç, Ankara/Turkey) was administered to provide sedation. Intravenous induction was performed with 2 mg/kg propofol (Propofol Lipuro 1% 200 mg/20 ml, B. Braun Medikal Dış Ticaret A.Ş., Esenler/Istanbul), 1 μg/kg fentanyl (Talinat ampoule 0.5 mg/10 ml, VEM İlaç San. ve Tic A.Ş, Çankaya/Ankara), and 6 mg/kg rocuronium (Esmeron® vial 50 mg/5 ml, Merck Sharp Dohme İlaçları Ltd. Şti., Levent/Istanbul). Female patients were intubated with 35Fr and male patients with 37Fr double-lumen endotracheal tubes (Teleflex Medical, Sheridan® Sher-i-Bronch® Endobronchial Tube). Fiberoptic bronchoscopy was used to confirm the correct placement of the endobronchial tube. After the intubation procedure, all patients underwent radial artery catheterization and subclavian central venous catheterization using a 3-lumen, 8.5F central venous catheter (Gemed Sağlık Ürünleri San. Tic. Ltd. Şti., Kartal/Istanbul).

During the perioperative period, a lung-protective mechanical ventilation strategy was employed during both double-lung ventilation and single-lung ventilation. Anesthesia maintenance was initiated with sevoflurane (Sevorane® Liquid 100%, Baxter Turkey Renal Services Inc., Ostim/Ankara) at a rate of 2 L/min in a mixture of 55% air and 45% oxygen, maintaining a minimum alveolar concentration (MAC) between 1.0 and 1.5. For intraoperative analgesia, remifentanil (Rentanil® vial containing 5 mg lyophilized powder, VEM İlaç San. ve Tic A.Ş, Çankaya/Ankara) was started at a dose of 0.15 mcg/kg/min. Throughout the operation, EtCO2 levels were maintained between 30-35 mmHg.

The ESPB OR TPVB procedures were performed while the patients were in the lateral position, after the completion of surgery, and before extubation. Sterile gloves were worn, and the puncture site was sterilized with 10% povidone-iodine in compliance with asepsis-antisepsis protocols. A fenestrated drape was placed, and the procedure was performed under ultrasound guidance (GE Logiq E ultrasound machine with a Linear IO 4-12 MHz probe, PENTA Elektronik Med. A.Ş, Ayrancı/Ankara) using the in-plane technique, An echoplex L 85 mm - 21G nerve block needle (85 mm, 21 gauge, Stimuplex® Ultra, B. Braun Melsungen AG, Hessen/Germany) was used for these procedures.

In Group 1, for ESPB, with the patient in the lateral position, a linear ultrasound probe (depth: 2-4 cm, frequency: 10-12 MHz) was used. After identifying the C7 spinous process by palpation, the probe was moved caudally to locate the T5 spinous process. The probe was placed parasagittally, 2-3 cm lateral to the spinous process. The T5 transverse process was visualized, and the block needle was advanced through the skin, passing through the trapezius, rhomboid, and erector spinae muscles until it contacted the transverse process (approximately 2-3 cm deep) using the in-plane technique. After confirming the absence of blood or air by negative aspiration and verifying the needle position by visualizing the needle tip and the injection of 1 mL of local anesthetic, a total of 20 mL of 0.5% bupivacaine (Buvasin 5 mg/mL vial, VEM İlaç, Çankaya/Ankara) was injected into the erector spinae plane. The distribution of the local anesthetic was observed in both cranial and caudal directions.

In Group 2, for TPVB, with the patient in the lateral position, a linear ultrasound probe (depth: 2-4 cm, frequency: 10-12 MHz) was used. After identifying the C7 spinous process by palpation, the probe was moved caudally to locate the T5 spinous process. The probe was placed parasagittally, 2-3 cm lateral to the spinous process. The trapezius, rhomboid major, and erector spinae muscles, along with the superior costotransverse ligament, were visualized from outer to inner structures. Clear ultrasound images of the pleura and T5 transverse process were obtained.

Using an in-plane technique, a block needle was advanced in a caudo-cranial direction, penetrating the superior costotransverse ligament. After confirming the absence of blood or air by negative aspiration, the position of the needle tip within the paravertebral space was verified by visualizing the needle tip and the injection of 1 mL of local anesthetic. Subsequently, a total of 20 mL of 0.5% bupivacaine (Buvasin 5 mg/mL vial, VEM İlaç, Çankaya/Ankara) was injected into the paravertebral space, and the downward displacement of the pleura was observed under ultrasound guidance.

All patients received a standard dose of IV 100 mg tramadol (Tramosel 100 mg/2 mL, Sandoz İlaç San. ve Tic. A.Ş., Kadıköy/Istanbul) 30-40 minutes before the end of the surgery. For nausea and vomiting prophylaxis, all cases were administered 10 mg metoclopramide (Anti-Nausea 10 mg/2 mL, Onfarma, Çankaya/Ankara), which has antiemetic and prokinetic effects, and the H2 receptor blocker ranitidine (Ranitab 50 mg/2 mL, Deva, Tuzla/Istanbul) during the intraoperative period.

At the end of the block procedures performed for postoperative analgesia, patients were decurarized with 2-4 mg/kg sugammadex (Bridion 200 mg/2 mL IV vial, Merck Sharp Dohme İlaçları Ltd. Şti., Levent/Istanbul). After extubation under appropriate conditions, they were transferred to the post-anesthesia care unit (PACU). Patients were monitored in the PACU for at least 30 minutes, and those with a Modified Aldrete Score of 9 or higher were transferred to the thoracic surgery intensive care unit (ICU) for close observation. For both groups, patients with an NRS score of 4-5 or a VAS score of 40-59 mm within the first 24 hours of evaluation received an additional IV 100 mg tramadol as analgesia. Patients with an NRS score ≥6 or a VAS score ≥60 mm were given 5 mg of subcutaneous morphine. No analgesics were administered to patients with an NRS score <4 or a VAS score <40 mm.

Patients who developed postoperative nausea and vomiting were treated with IV 10 mg antiemetic. Those who experienced pruritus were administered IV 20 mg prednisolone (methylprednisolone 20 mg/lyophilized ampoule, Gensenta İlaç Sanayi ve Ticaret A.Ş., Beşiktaş/Istanbul) along with IV antihistamine (pheniramine maleate 45.5 mg/2 mL, Sandoz İlaç San. ve Tic. A.Ş., Kadıköy/Istanbul).

Statistical Analysis Descriptive statistics of the data obtained from the study are presented as the mean and standard deviation for numerical variables and frequency and percentage analysis for categorical variables. Independent samples t-test and Chi-square test were used to compare demographic characteristics between study groups. Additionally, repeated measures analysis of variance (ANOVA) was used to compare numerical variables measured at different time points across the study groups. Analyses were performed using the SPSS 22.0 software, with a significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone thoracotomy, with ASA I,II,III physical status and received ESP block or paravertebral block

Exclusion Criteria:

* Patients were excluded from the study if they were emergency cases, had an ASA class IV or V status, had peripheral vascular disease, were pregnant, had heart failure, were allergic to local anesthetics, or if their medical records were inaccessible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Postoperative 0., 3., 6., 12., ve 24. hour
  Visual analog scale, is one of the pain rating scales, providing a range of scores from 0-100.

SECONDARY OUTCOMES:
side effects | Postoperative 24 hours
  Side effects including postopertive nausea, pruritus and shoulder pain

CONTACTS AND LOCATIONS:
Overall Officials: Elzem Sen, Assoc. Prof, Study Director — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No